| 1 | |
|---|---|
| 2 | |
| 3 | |
| 4<br>5 | EFFICACY OF GABAPENTIN FOR POST-COVID-19 OLFACTORY DYSFUNCTION |
| 6 | |
| 7 | |
| 8 | Principal Investigator: Jay Piccirillo, MD, Department of Otolaryngology-Head and Neck Surgery |
| 10 | |
| 11 | |
| 12 | |
| 13 | |
| 14 | |
| 15 | |
| 16 | |
| 17 | |
| 18 | Version Date/Number: |
| 19 | 06/20/22,V11 |
| 20 | |
| 21 | |
| 22 | |
| 23 | |

# TABLE OF CONTENTS

| 26 | A IN | TRODUCTION | 4 |
|----|-------------|-------------------------------------------------|----|
| 27 | A1 | STUDY ABSTRACT | 4 |
| 28 | A2 | PRIMARY HYPOTHESIS | |
| 29 | A3 | PURPOSE OF THE STUDY PROTOCOL | |
| 30 | B BA | ACKGROUND | 4 |
| 31 | B1 | Prior Literature and Studies | 5 |
| 32 | B2 | RATIONALE FOR THIS STUDY | 6 |
| 33 | C ST | UDY OBJECTIVES | 6 |
| 34 | C1 | Primary Aim | 6 |
| 35 | C2 | SECONDARY AIM | 6 |
| 36 | C3 | RATIONALE FOR THE SELECTION OF OUTCOME MEASURES | 6 |
| 37 | D IN | VESTIGATIONAL AGENT | 8 |
| 38 | D1 | Preclinical Data | 8 |
| 39 | D1 | CLINICAL DATA TO DATE | |
| 40 | D3 | Dose Rationale and Risk/Benefits | |
| 41 | 20 | UDY DESIGN | _ |
| 42 | E1 | OVERVIEW OR DESIGN SUMMARY | |
| 43 | E2 | SUBJECT SELECTION AND WITHDRAWAL | |
| 44 | 2.a | = | |
| 45 | 2.a | | |
| 46 | 2.b | = | |
| 47 | 2.0 | J | |
| 48 | 2.a | | |
| 49 | 2.e | J | |
| 50 | 2.f | | |
| 51 | 2.g | | |
| 52 | 2.h | 1 0 | |
| 53 | E3 | Study Drug | |
| 54 | 3.a | T | |
| 55 | 3.b | = | |
| 56 | 3.0 | | |
| 57 | 3.a | · | |
| 58 | 3.e | J | |
| 59 | 3.f | 1. | |
| 60 | 3.g | | |
| 61 | 3.h | | |
| 62 | 3. <i>i</i> | Receiving, Storage, Dispensing and Return | 14 |
| 63 | F ST | UDY PROCEDURES | 14 |
| 64 | | Screening for Eligibility | |
| 65 | | SCHEDULE OF MEASUREMENTS | |
| 66 | F3 | SAFETY AND ADVERSE EVENTS | |
| 67 | 3.a | <i>y y</i> 1 | |
| 68 | 3.a | 8 | |
| 69 | | i Investigator only | |
| 70 | <i>3.b</i> | Definitions of Adverse Events | 18 |

| 71 | i Relationship | |
|----------|-------------------------------------------------|----|
| 72<br>73 | ii Severity | |
| 73<br>74 | iii Expectedness | |
| 75 | 3.d Reporting Procedures | |
| 76 | 3.e Adverse Event Reporting Period | |
| 77 | F4 STUDY OUTCOME MEASUREMENTS AND ASCERTAINMENT | |
| 78 | G STATISTICAL PLAN | 21 |
| 79 | G1 SAMPLE SIZE DETERMINATION AND POWER | 21 |
| 80 | G2 INTERIM MONITORING AND EARLY STOPPING | 21 |
| 81 | G3 STATISTICAL METHODS | |
| 82 | G4 MISSING OUTCOME DATA | |
| 83 | G5 Unblinding Procedures | 22 |
| 84 | H DATA HANDLING AND RECORD KEEPING | |
| 85 | H1 CONFIDENTIALITY AND SECURITY | |
| 86 | H2 RECORDS RETENTION | 23 |
| 87 | I STUDY ADMINISTRATION | 23 |
| 88 | I1 SUBJECT STIPENDS OR PAYMENTS | 23 |
| 89 | I2 Study Timetable | |
| 90 | J PUBLICATION PLAN | 23 |
| 91 | K ATTACHMENTS | 23 |
| 92 | K1 QUESTIONNAIRES OR SURVEYS | 23 |
| 93 | L REFERENCES | 24 |
| 0.4 | | |
| 94 | | |
| 95 | | |
| ,, | | |
| 96 | | |
| 97 | | |
| 98 | | |
| 99 | | |
| ,, | | |
| 100 | | |
| 101 | | |
| 102 | | |
| 102 | | |
| 103 | | |
| 104 | | |

#### **A** Introduction

106107

108

## A1 Study Abstract

olfactory dysfunction.

109 COVID-19 has now infected over 33 million people in the United States and approximately 185 million worldwide. 1,2 Of those, an estimated 85% have reported either 110 111 a new clinical diagnosis or subjective onset of olfactory dysfunction.<sup>3</sup> While most patients will recover their sense of smell within 7-14 days, others may not return to their 112 113 baseline function for months or at all. Viral infections that target the upper respiratory 114 system, such as COVID-19, often leave patients with diminished olfaction. This new-115 onset anosmia, hyposmia, and parosmia is theorized to be caused by damage to sensory 116 neurons following viral insult. Unfortunately, there is no treatment for post-COVID 117 olfactory dysfunction. Most patients are recommended to perform olfactory training with essential oils, but the evidence base to support this recommendation is not firm. Thus, 118 119 there is a very big need for effective treatments for patients suffering from post-COVID

120 121 122

123

124

125

126

127

128

129 130

131

One potential therapy is gabapentin. Used as an antiepileptic and now first-line medication for the treatment of diabetic neuropathy, gabapentin is known for reducing pain secondary to diabetic neuropathy and post-herpetic neuralgia. Gabapentin works mainly on voltage-gated calcium channels (VGCC) with an ability to cross the basement membrane, a trait important for an antiepileptic. The  $\alpha2\delta2$  subunit of VGCCs, with increased expression in corticospinal neurons, has been associated with loss of regrowth after spinal injuries. The  $\alpha2\delta2$  blockage by gabapentin can allow increased nerve regeneration and return of function. Inhibition of the  $\alpha2\delta2$  subunit on VGCCs may allow nerves to regenerate more rapidly than physiologically normal. This study will evaluate the efficacy of gabapentin for olfactory dysfunction (anosmia, hyposmia, parosmia) in

post-COVID-19 patients.

# 133 A2 Primary Hypothesis

- We hypothesize that oral gabapentin will be more effective than placebo for COVID-19-
- related olfactory dysfunction (OD) improvement.

# 136 A3 Purpose of the Study Protocol

- 137 This study will evaluate the efficacy of gabapentin for olfactory dysfunction (anosmia,
- 138 hyposmia, parosmia) in post-COVID-19 patients.

139

# B Background

### B1 Prior Literature and Studies

The SARS-CoV-2 virus, has infected an estimated 78 million in the United States with ~85% of patients reporting some form of olfactory dysfunction. <sup>1,3</sup> More recent studies have shown an increased prevalence of olfactory change reported in women over men and in Western countries when compared to Eastern countries. <sup>8,9</sup> Moreover, the percentage of patients with post-COVID-19 olfactory dysfunction is thought to be underreported as patients need to individually report the symptom to their physician for it to be recorded. <sup>9</sup>

Evidence has emerged to explain the pathophysiology of COVID-19 and its mechanism of action on neurosensory pathways. Research suggests that COVID-19 affects two genes commonly found in the human respiratory system, ACE2 and TMPRSS2.<sup>10</sup>. ACE2, commonly associated with the renin-angiotensin-aldosterone system, has another role as a receptor protein on cell surfaces – a receptor proven vital for SARS-CoV-2 to enter respiratory cells. 11 Similarly, TMPRSS2 also plays a role in SARS-CoV-2 entry into cells and both genes are expressed in neuronal support cells. ACE2 and TMPRSS2 are found only in support cells and not neurons. The support cells, such as sustentacular cells, degenerate and are unable to sustain neurons. This lack of neuronal stability is what likely causes the temporary neurosensory loss seen in post-COVID-19 patients. However, evidence is now also supporting the theory that COVID-19-related olfactory dysfunction may be due to direct damage to olfactory receptor neurons (ORNs) as well, which would increase recovery time as neurons regenerate more slowly. Previous strains of human coronavirus have also been proven to target ORNs causing olfactory dysfunction but whether this direct damage to neurons is related to ACE2 and TMPRSS2 has yet to be determined.<sup>10</sup>

Patients who do recover their sense of smell after infection tend to notice improvement in just weeks, paralleling the rapid recovery rate of support cells. Those with lingering olfactory dysfunction either return to new normalcy in months instead of weeks or have yet to return to baseline. Some patients report a return of smell followed shortly by new smell distortion. This observation of differing recovery rates supports the theory that SARS-CoV-2 also damages olfactory receptor neurons directly leading to longer recovery times. Research has demonstrated the possible utility in olfactory training, a therapy thought to encourage neuroplasticity via repeat exposure to odors. However, the evidence to support this treatment is not universally accepted and pharmacotherapy options for post-COVID-19 olfactory dysfunction are still being explored; one potential therapy is gabapentin.

Gabapentin is an antiepileptic medication now used as first-line therapy for diabetic neuropathy and herpetic neuralgia. Gabapentin works by binding to VGCCs, which play an important role in neuronal synaptic transmission. More specifically, gabapentin binds to  $\alpha_2\delta$  isoforms which have been associated with neuropathic pain. The postsynaptic  $\alpha_2\delta 1$  subunit promotes spinogenesis, the development of neuronal dendritic spines, while the  $\alpha_2\delta 2$  works as a suppressor of axonal regeneration. <sup>13</sup> Gabapentin functions as an inhibitor of the  $\alpha_2\delta 2$  subunit and therefore blocks the suppression of axonal regeneration leading to increased neuronal regeneration and function. The medication is effective in the treatment

188 of chronic pain and burning mouth syndrome (BMS). The mode of action is thought to be 189 primarily due to the fact that gabapentin is highly lipophilic and can enter the central nervous system (CNS) and iad in neuron regeneration. <sup>14</sup> For these reasons, gabapentin is 190 191 thought to have the potential to improve post-COVID-19 olfactory dysfunction caused by 192 neuronal damage. Our study will investigate the efficacy of gabapentin to increase 193 recovery of olfactory dysfunction secondary to post-COVID-19 infection. 194 195

#### B2Rationale for this Study

196 Olfactory dysfunction is a major symptom of SARS-CoV-2 affecting up to 80% of 197 infected individuals. While most have a return to normal olfactory function in weeks, 198 some may not see full improvement for months and a small percentage may not recover 199 function and suffer long-term physical limitation and functional impairment. This 200 placebo-controlled, double-blinded pilot RCT will evaluate the efficacy of oral 201 gabapentin to improve chronic (>3 months) olfactory dysfunction secondary to COVID-202 19 infection. This study will provide data on the efficacy of gabapentin for the treatment 203 of OD.

204

# **Study Objectives**

205 206

#### 207 *C1* Primary Aim

- 208 To evaluate the efficacy of oral gabapentin on improvement of olfactory dysfunction in 209 patients with post-COVID-19 anosmia, hyposmia, or parosmia. Participants will receive a 210 maximum of 14weeks of either gabapentin or placebo with the first four weeks serving as
- 211 a titration phase and the last two weeks serving as a taper-down period.

#### 212 *C2* Secondary Aim

213 Describe the adverse effects of gabapentin. All participants will be monitored for adverse 214 effects throughout the study.

# Rationale for the Selection of Outcome Measures

216 217

215

### Primary Outcome:

218 Clinical Global Impression of Improvement Scale (CGI-I). The response rate is 219 defined as the number of participants self-reporting minimal change or larger on 220 the Clinical Global Impression of Improvement Scale (CGI-I) scale, divided by 221 the number of participants in each group. The CGI-Improvement is a self-222 reported scale of improvement ranging from 1 to 7 (1 is Very Much Improved, 7 223 is Very Much Worsened) and will be measured after completing 8 weeks of the 224 fixed, highest-tolerable dose. Each rating is well defined to maximize accuracy. 225 Participants reporting 3 as Minimally Improved, 2 as Much Improved, or 1 as Very 226 Much Improved in the CGI-I will be deemed responders to treatment, and the 227 number of responders to non-responders will be compared between the two arms -228 CGI-Severity (CGI-S) and CGI-Improvement (CGI-I).

231

# **Secondary Outcomes:**

- 232 233 234
- 235 236
- 237 238 239
- 241 242 243

240

- 244 245
- 246 247
- 248 249
- 250

- 1. **CGI-Severity.** The *CGI-Severity* scale ranges from 1 to 7, where 1 is normal function and 7 is complete anosmia. This assessment will provide subjective data on patients' baseline olfactory function prior to beginning the trial, after 8-week Fixed-Dose period, and 4 weeks after completion of Taper-Down phase.
- 2. **CGI-Improvement**. The CGI Improvement will also be administered 4 weeks after completion of Taper-Down phase which same analysis as described above.
- 3. University of Pennsylvania Smell Identification Test (UPSIT). 15 The UPSIT is composed of 40 strips of microencapsulated odorants, which are present on the bottom of each page, just below a four-alternative multiple-choice question. For a given item, the patient releases an odor by scratching the microencapsulated pad with a pencil tip, smells the pad, and indicates the odor quality from four alternatives. Even if no smell is perceived, a response is required (i.e., the test is forced-choice). The subject's total correct score out of the 40 items is determined.<sup>16</sup>

The total UPSIT score can range from 0 to 40 and scores are interpreted as the level of absolute smell function (i.e., normosmia, mild hyposmia, moderate hyposmia, severe hyposmia, and anosmia), using the age- and sex-related normative classification system described in the UPSIT manual (Table 1) The minimal clinically important difference in UPSIT score is 4.

| Disease Classification | | | |
|------------------------|----------|-------------|-------|
| Based on UPSIT | | Women | Men |
| Normosmia | | >34 | >33 |
| Hyposmia | | | |
| | Mild | 31-34 | 30-33 |
| | Moderate | 26-30 | 26-29 |
| | Severe | 19-25 | |
| Anosmia | | 6-18<br>≤ 5 | |
| Malingering | | | |

253 254

251 252

- 255 256 257
- 259 260 261 262

- 263 264 265
- 266 267 268 269

- 4. Olfactory Dysfunction Outcomes Rating (ODOR). The ODOR questionnaire is a 28-item disease-specific health status survey to assess the physical problems, functional impairments, and emotional consequences secondary to olfactory dysfunction. ODOR was developed and validated by Dr. Jake Lee and colleagues in the Clinical Outcomes Research Office at Washington University.
- **5.** NASAL-7. NASAL-7 is a simple diagnostic tool for olfactory dysfunction that is based on commonly found household items and can be used by adults who suspect olfactory dysfunction. The NASAL-7 was developed by Dr. Piccirillo and colleagues in the Clinical Outcomes Research Office. The NASAL-7, contains 7 household items with each item scored as 0 for 'Cannot Smell', 1 for 'Smells Less Strong/Different Than Normal', and 2 for 'Smells Normal', for a total possible score ranging from 0-14. The following four categories of olfactory function were defined based on NASAL-7 score: anosmia (score 0-4), severe dysfunction (score 5-7), mild dysfunction (score 8-10), and normosmia (score 11-14).
- 6. Clinical Global Impression-Severity Scale for Parosmics (CGI-P). The CGI-P Scale is a global rating of parosmia and the single global rating ranges from 1-5, where 1 is No Distortion, 2 is Mild Distortion, 3 is Moderate Distortion, 4 is Mostly Distorted, and 5 is Complete Distortion. The response on the CGI-P will

270 provide information on the patient's perceived severity of the distortion of their 271 smell. 272 273 D **Investigational Agent** 274 275 Preclinical Data **D**1 276 Gabapentin is an antiepileptic medication now used as first-line therapy for diabetic 277 neuropathy and herpetic neuralgia. Gabapentin works by binding to voltage-gated 278 calcium channels (VGCCs), which play an important role in neuronal synaptic 279 transmission. More specifically, gabapentin binds to  $\alpha_2\delta$  isoforms which have been 280 associated with neuropathic pain. 281 282 The  $\alpha 2\delta 2$  subunit of VGCCs, with increased expression in corticospinal neurons, has 283 been associated with loss of regrowth after spinal injuries. The postsynaptic  $\alpha_2\delta 1$  subunit 284 promotes spinogenesis, the development of neuronal dendritic spines, while the  $\alpha_2\delta_2$ works as a suppressor of axonal regeneration. The  $\alpha 2\delta 2$  blockage by gabapentin can 285 allow increased nerve regeneration and return of function. <sup>7</sup> Inhibition of the α2δ2 subunit 286 287 on VGCCs may allow nerves to regenerate more rapidly than physiologically normal. 288 Clinical Data to Date D2289 Gabapentin is an antiepileptic medication now used as first-line therapy for diabetic 290 neuropathy and herpetic neuralgia. Gabapentin works by binding to voltage-gated 291 calcium channels (VGCCs), which play an important role in neuronal synaptic 292 transmission. More specifically, gabapentin binds to  $\alpha_2\delta$  isoforms which have been 293 associated with neuropathic pain. 294 295 The medication has also proven effective in treated chronic pain from Burning Mouth 296 Syndrome (BMS) since gabapentin is highly lipophilic and can enter the central nervous 297 system (CNS). <sup>14</sup> For these reasons, gabapentin is thought to have the potential to improve post-COVID-19 olfactory dysfunction caused by neuronal damage. Gabapentin can 298 299 penetrate the blood-brain barrier and enter the CNS where it can aid in neuron 300 regeneration. 301 Dose Rationale and Risk/Benefits D3302 Gabapentin dosing for this study mirrors dosing for the prior study "Relief of Idiopathic 303 Subjective Tinnitus" (IRB #02-0717) 304 Following randomization, participants in the gabapentin arm will take gradually titrated 305 dosages in order to achieve a dose of 3600mg/d or highest tolerable dose. The titration 306 schedule will span a maximum 4 weeks to reach 3600mg/d. 307 Week 1, 900 mg/d Week 2, 1800 mg/d 308 309 Week 3, 2700 mg/d 310 Week 4, 3600 mg/d 311

Gabapentin (300 mg per capsule) and placebo will be supplied to patients in identical opaque capsules in blinded fashion. The medications will be distributed in 4 separate vials representing each of the four weeks of the Titration Period. All participants will be provided an equal number of capsules and instructed to follow a TID (i.e., 3 times per day) dosing schedule. All participants' dosages will be titrated to a maximum dose of 3600 mg/d, regardless of any possible beneficial effect achieved at lower dosages. If intolerable adverse reactions occur, the dosage will be decreased to previous tolerable dose (e.g. if 2700mg/d is intolerable, dosage will be decreased to 1800 mg/d). If, during the first week, 900 mg/d is intolerable, dosing will be decreased by 300 mg/d per day until tolerable (i.e., 600 mg/d, 300mg/d) or until they are no longer taking the medication. The dose established during the Titration Period will be maintained throughout the Fixed-Dose period. Participants receiving the matching placebo capsules will be provided similar instructions for titration and de-escalation, should side effects develop.

The potential benefit to the participant is improvement of their olfactory dysfunction using this therapy. The potential benefit to the society is the use of the pilot study results to initiate a larger trial to further evaluate the efficacy of gabapentin in the treatment of post-COVID-19 olfactory dysfunction.

The potential risk to participants during the study is an adverse event associated with the medication use. Abrupt cessation of gabapentin may alter the seizure threshold; for this reason, participants will be provided with a taper schedule specific to the gabapentin dose at time of completion of the Fixed Dose period. Gabapentin has a slight risk of dependence in patients with previous history of alcohol, cocaine, or opioid abuse so these individuals will be excluded from the study. <sup>17</sup>

## E Study Design

### E1 Overview or Design Summary

This study will be a double-blinded, placebo-controlled, randomized pilot clinical trial to evaluate the efficacy of gabapentin to improve post-COVID-19 olfactory dysfunction.

This study will also describe adverse effects related to oral gabapentin use.

This study will be conducted via virtual research guidelines and procedures. We will not require in-person patient participation or evaluation. Following initial evaluation to ensure potential participants meet all inclusion criteria and none of the exclusion criteria, the research study will be explained in full via Zoom call, phone call if necessary. Participants will then be randomized in a 1:1 allocation via permuted-block sequencing into the oral gabapentin group or the placebo group. All assessments will be conducted through a HIPAA-compliant online survey form. Baseline assessments will help us determine subjective and objective rates of olfactory dysfunction. Assessments will be conducted again after the 8-week Fixed-Dose period and 4 weeks after completing taper.

The primary objective of this study is to assess the efficacy of oral gabapentin in 355 356 improving olfactory dysfunction secondary to COVID-19. 357 E2Subject Selection and Withdrawal 358 359 2.a **Inclusion Criteria** 360 Participants will be recruited based on the following inclusion criteria: 361 Men and women between the ages of 18 and 65 years 362 Residing within the states of Missouri or Illinois 363 Clinically diagnosed or subjective olfactory dysfunction (anosmia, hyposmia, 364 or parosmia) of at least 3 months duration associated with COVID-19 365 infection 366 initial UPSIT score consistent with diminished olfactory function (score > 6 367 and  $\leq 33$  in men and score > 6 and  $\leq 34$  in women). Willing to respond daily to study surveys, preferably through smartphone with 368 unlimited texting plan. 369 370 In possession of all 7 household items associated with NASAL-7: soap, burnt 371 candle, peanut butter, herb, garlic, lemon, and coffee 372 373 2.a **Exclusion Criteria** 374 Individuals will not be allowed to participate in this study if they meet one or more of the 375 following exclusion criteria: 376 Clinically diagnosed olfactory dysfunction secondary to non-COVID-19 viral 377 infection, genetic abnormalities or congenital dysfunction, trauma, nasal 378 polyps, neurodegenerative disorders 379 Current use of: azelastine, bromperidol, orophenadrine, oxomemazine, 380 kratom, paraldehyde, or thalidomide 381 History of addiction to alcohol, cocaine, or opioids 382 Impaired renal function, myasthenia gravis, or myoclonus 383 Severe allergy to peanuts Pregnancy or attempting pregnancy during study participation 384 385 Inability to participate in virtual trial due to lack of access to the; inability to 386 comprehend or use English language Availability less than 18 weeks from time of enrollment 387 Residency in states other than Missouri or Illinois. 388 389 **2.b Ethical Considerations** 390 This study relies on participation of human subjects. Informed consent will be 391 obtained from each participant to ensure their safety, minimize risk, and ensure full 392 confidentiality. All assessments will be conducted virtually via HIPAA-compliant online 393 surveys at baseline and then throughout the study course. Selection of participants for the 394 study will consider the variability in response to COVID-19 as well as response to 395 gabapentin by ensuring the two groups are matched 1:1 by permuted block 396 randomization. Gabapentin has a slight risk of dependence in individuals with previous

\_\_\_\_\_

- 397 history of alcohol, cocaine, or opioid abuse so these patients will be excluded from the
- 398 study. <sup>17</sup>The study team will be available at all times for participants during the full course
- 399 of the trial.

400

# 2.c Subject Recruitment Plans and Consent Process

- 401 Recruitment will be done at the Washington University Department of Otolaryngology-
- Head and Neck Surgery outpatient clinics. Advertisements will also be sent to all
- 403 members of the St. Louis ENT Club, and otolaryngologists whose practices are within
- 404 150 miles of Washington University Medical Center (WUMC). Direct recruitment of
- potential participants will also be achieved through use of the Washington University
- 406 Volunteers for Health Research Participant Registry, and the Otolaryngology Research
- 407 Participant Registry. This recruitment strategy has been successful for two current trials
- 408 of treatment for COVID-associated anosmia VOLT (IRB ID# 202011046) and SCENT2
- 409 (IRB ID# 202101190). We may also attempt to recruit potential participants from past
- studies in our lab, such as the CODS trial (IRB ID# 202004146). Additionally, due to the
- focus on virtual research at this time, we may also use website postings and work with
- anosmia support groups such as AbScent and FifthSense to share the trial.

### 413 2.d Randomization Method and Blinding

- Participants who remain eligible at the end of the screening period will be randomized in
- a double-blind fashion, according to a computer-generated random code, to receive either
- 416 placebo or gabapentin. Dr. Kallogieri will provide the randomization table to the BJH
- Research Pharmacist, who will prepare both gabapentin and placebo for the entire study.
- The research assistants will collect the gabapentin and placebo in a blinded fashion from
- 419 the research pharmacist for distribution to the participants via FedEx.

## 420 **2.e** Risks and Benefits

- The potential benefit to the participant is improvement of their olfactory dysfunction
- 422 using this therapy. The potential benefit to the society is the use of the pilot study results
- 423 to initiate a larger trial to further evaluate the efficacy of gabapentin in the treatment of
- 424 post-COVID-19 olfactory dysfunction.

425

- The potential risk to participants during the study is an adverse event associated with the
- 427 medication use. Abrupt cessation of gabapentin may alter the seizure threshold; for this
- reason, participants will be provided with a taper schedule specific to the gabapentin dose
- at time of cessation. Gabapentin has a slight risk of dependence in individuals with
- previous history of alcohol, cocaine, or opioid abuse so these individuals will be excluded
- 431 from the study. <sup>17</sup>

432

- The consent process informs a volunteer about the study, indicates that participation is
- voluntary, and that he/she has the right to stop at any time. Risks are listed in the
- informed consent form and described orally during the consent process.

| 437 | 2.f Early Withdrawal of Subjects |
|---|---|
| 438 | If a subject decides to withdraw from all components of the research study, the |
| 439 | investigator will discontinue all of the current and scheduled research activities in the |
| 440 | study. Participants taking an intervention medication at the time of withdrawal will be |
| 441 | provided with a taper-down schedule based on maximum intervention dose achieved. |
| 442 | provided with a taper-down schedule based on maximum mer vention dose demoved. |
| TT <u>L</u> | |
| 443 | 2.g When and How to Withdraw Subjects |
| 444 | A participant can withdraw consent for the study at any time. Participants will be allowed |
| 445 | to end participation in the study at any point should they desire. If a participant must be |
| 446 | withdrawn due to a drug-related serious adverse event, then blind will be broken and, if |
| 447 | on gabapentin, drug withdrawal will be tapered or completely stopped based on the |
| 448 | clinical judgement of the PI. All participants will have an exit interview to ascertain any |
| 449 | adverse effects and discuss the reason for ending participation. The study team will |
| 450 | follow them for safety reasons up to 30 days after stopping use of the study drug. |
| 451 | |
| 452 | 2.h Data Collection and Follow-up for Withdrawn Subjects |
| 453 | If a participant has ended participation, the only data that will be collected are the data |
| 454 | from the exit interview and the data collected prior to withdrawal. There will not be any |
| 455 | other follow-up or data collected from these subjects. |
| 456 | other renew up of data confected from these subjects. |
| 457 | Data collected up to this point will not be used in the analysis, and further data will not be |
| 458 | collected from these participants. |
| 459 | conceted from these participants. |
| 460 | E3 Study Drug |
| 461 | Lo Study Drug |
| +01 | |
| 462 | 3.a Description |
| 463 | Gabapentin is an antiepileptic medication now used as first-line therapy for diabetic |
| 464 | neuropathy and herpetic neuralgia. Gabapentin works by binding to voltage-gated |
| 465 | calcium channels (VGCCs), which play an important role in neuronal synaptic |
| 466 | transmission. More specifically, gabapentin binds to $\alpha_2\delta$ isoforms which have been |
| 467 | associated with neuropathic pain. |
| 468 | 3.b Treatment Regimen |
| 469 | During the titration period of maximum 4 weeks, participants randomized to |
| 470 | the gabapentin arm will take gradually titrated dosages of gabapentin as follows: |
| 471 | Week 1, 900 mg/d (300 mg TID) |
| 472 | Week 2, 1800 mg/d (600 mg TID) |
| 473 | Week 3, 2700 mg/d (900 mg TID) |
| 474 | Week 4, 3600 mg/d (1200 mg TID) |
| 475 | (1200 mg 112) |
| 476 | If intolerable effects occur, dosage will be decreased by 1 dose (300 mg) step (e.g. if |
| 477 | 2700 mg/d is intolerable, dosage will be decreased to 2400 mg/d). Further de-escalation |

- will be determined by PI clinical judgement to prior tolerable dose. The highest tolerable
- dose established during the Titration Period will be maintained throughout the 8-week
- 480 Fixed-Dose period.

# 481 3.c Method for Assigning Subjects to Treatment Groups

- The participants will be divided using permuted block randomization in a 1:1 allocation
- between two arms: the oral gabapentin group and the oral lactose placebo group with 20
- persons in each group.

# 485 3.d Preparation and Administration of Study Drug

- Gabapentin (300 mg per capsule) and placebo will be supplied to patients in identical
- opaque capsules in blinded fashion. The medications will be distributed in 4 separate
- vials representing each of the four weeks of the Titration Period and distributed in 8
- separate vials prior to the Fixed-Dose period.

# 490 3.e Subject Compliance Monitoring

- There will be check-ins with the study participants every two weeks conducted virtually
- through the participant's preferred communication method (i.e. phone call or video call)
- 493 to answer questions and ensure participants are adhering to medication schedule. Subjects
- will be asked to keep a paper calendar for daily notes of pill count, side/adverse effects,
- and study barriers. The paper calendar will be mailed back to the RA after study
- 496 completion.

# 497 3.f Prior and Concomitant Therapy

- 498 Patients receiving concomitant therapy specifically for the treatment of olfactory
- dysfunction will not be eligible for the trial unless they are able to stop taking those
- therapies during the conduct of the study. Participants who have tried previous therapies
- for their olfactory dysfunction, including over-the-counter treatments such as vitamin A
- or omega-3 fatty acids will be eligible for the trial. Information will be gathered on their
- use of prior or current therapies, and if needed, a sensitivity or subgroup analysis may be
- 504 considered.

# 505

506

509

### 3.g Packaging

- The Research Pharmacist will deliver the gabapentin and placebo in a blinded fashion to
- 508 the research assistant for distribution to the participants via FedEx.

### 3.h Blinding of Study Drug

- Participants will be divided into two groups; one group will be given oral gabapentin
- while the other group will be given oral placebo. The research pharmacist will receive the
- randomization assignment code from the biostatistician. The RA will pick up the study
- drug in blinded fashion from research pharmacist and distribute it to the participant via
- FedEx delivery. In this way, only the Research Pharmacist will know participant
- assignment. Adequate taper of gabapentin will be provided for those on gabapentin while
- 516 the placebo group will receive additional placebo for taper in order to maintain the blind.

#### 3.i Receiving, Storage, Dispensing and Return

- 518 The services of the Investigational Pharmacy at Barnes-Jewish Hospital will be used for
- 519 this trial. The product used in this trial will be managed by the pharmacist according to
- 520 the pharmacy SOP.

### **Study Procedures**

521 522

523

528 529

533

535

536

537

538

539

517

#### **F1** Screening for Eligibility

524 Individuals who reach out with interest in the study after seeing the approved study flyer

or who have contacted RA for participation in similar studies for which recruitment has 525 526

ended will asked to complete an online screening questionnaire (survey titled:

527 "ScreeningSurvey") to ensure he or she meets all the inclusion criteria and does not meet

any exclusion criteria. Following eligibility confirmation, the RA will collect information

required to mail screening smell identification test (UPSIT). Once received, the

530 participant will complete the UPSIT and provide their response virtually through the

531 REDCap survey. Once eligibility is confirmed based on UPSIT score, participants will

532 be provided through REDCap an online consent form to review and complete. The RA

will offer each participant the option to review the consent form independently or with

the RA via zoom or phone call (zoom as the preferred option). Once the participant 534

electronically signs the consent form, the RA will review it and sign. The REDCap

software will automatically email the participant a copy of their completed form.

#### F2Schedule of Measurements

Following the recruitment period and successful enrollment, baseline survey completion

(survey titled Week0BaselineSurvey) and randomization of participants will occur. The

timeline for measurements can be seen below.

540 541 542

543 544

545

546

547

548

### **Gabapentin Study Flow Chart**



| 49 | |
|---|---|
| 50 | |
| 51 | |
| 2 | |
| 3 | |
| 4<br>5<br>6<br>7 | a. Federal guidelines require timely reporting (within 15 calendar days) of an unanticipated or life-threatening event or death occurring within 30 days of active study participation. |
| 58<br>59 | Titration Period: maximum duration 4 weeks |
| 0 | THE |
| 1 | Placebo. In this study, we plan to use an inert placebo and not an active drug |
| 2 | or non-active drug with side effects similar to gabapentin. Participants randomized to the |
| 3 | Placebo arm will participate in a 4-week Titration Period. Placebo will be supplied to |
| | patients in opaque capsules in blinded fashion. The medications will be distributed in 4 |
| | separate vials representing each of the four weeks of the Titration Period. If intolerable |
| | adverse reactions occur, the dosage will be decreased to prior tolerable dose. |
| | Gabapentin. Participants randomized to the gabapentin arm will take gradually titrated dosages of gabapentin as follows: |
| | gradually thrated dosages of gaoapentili as follows. |
| | Week 1, 900 mg/d (300 mg TID) |
| | Week 2, 1800 mg/d (600 mg TID) |
| | Week 3, 2700 mg/d (900 mg TID) |
| | Week 4, 3600 mg/d (1200 mg TID) |
| | Gabapentin (300 mg per capsule) will be supplied to participants in opaque |
| | capsules in blinded fashion identical to the supply of Placebo. The medications will be |
| | distributed in 4 separate vials representing each of the four weeks of the Titration Period. |
| | All participants' dosages will be titrated to a maximum dose of 3600 mg/d, regardless of |
| | any effect achieved at lower dosages. If intolerable effects occur, dosage will be |
| | decreased by 1 dose (300 mg) step (e. g. if 2700 mg/d is intolerable, dosage will be |
| | decreased to 2400 mg/d). Further de-escalation will be determined by PI clinical |
| | judgement to prior tolerable dose. Participants with intolerable effects may have a lower |
| | maximum dose than 3600mg/d and may complete the Titration Period in less than 4 |
| 1 | weeks. The dose established during the Titration Period will be maintained throughout |

the Fixed-Dose period.

| WEEK 1 | WEEK 2 | WEEK 3 | WEEK 4 |
|---|---|---|---|
| 900 MG | 1800 MG | 2700 MG | 3600 MG |
| 1 MORNING<br>1 NOON<br>1 NIGHT<br>(21 PILLS) | 2 MORNING<br>2 NOON<br>2 NIGHT<br>(42 PILLS) | 3 MORNING<br>3 NOON<br>3 NIGHT<br>(63 PILLS) | 4 MORNING<br>4 NOON<br>4 NIGHT<br>(84 PILLS) |

Gabapentin (300 mg pill) Titration Schedule

If at any point during the Titration Period, the participant wishes to discontinue the medication for any reason, they will be instructed to follow the taper down schedule (see below) in order to safely stop the medication. The participant will be informed that any abrupt stoppage of gabapentin could cause serious adverse effects.

Participants will be contacted by telephone or video call by the Research Assistant (RA) at the end of Titration period. The purpose of this call will be to query the participants about adverse effects. Participants will be provided with a paper calendar and asked to maintain diaries of olfactory and taste symptoms and adverse effects possibly related to the intervention.

Participants will not complete any forms at the completion of Titration period. Instead, they will proceed directly to Fixed-Dose Period.

### Fixed-Dose Period: duration 8 weeks

During the Fixed-Dose period, participant's dose will remain at their maximum tolerated dosage established during the Titration phase. The study drug will be distributed in eight separate vials representing the eight weeks of the Fixed-Dose period. The RA will contact the participants at the end of Week 4 to administer the blind assessment using REDCap (survey titled: "Blind Assessment"). Participants will complete the following forms after completing the Fixed-Dose Period (survey titled: "FixedDoseSurvey"):

- 1.) Clinical Global Impression of Severity Scale (CGI-S).
- 2.) Clinical Global Impression of Improvement Scale (CGI-I)
- 3.) University of Pennsylvania Smell Identification Test (UPSIT)
- 4.) Olfactory Dysfunction Outcomes Rating (ODOR)
- 5.) *NASAL-7*
- 6.) Clinical Global Impression-Severity Scale for Parosmics (CGI-P)
- 7.) Adverse Event assessment
- 8.) Compliance

Adverse events. Any unintentional or unfavorable clinical sign or symptom, any new illness or disease or the deterioration of existing disease or illness, or any clinically significant deterioration in any laboratory assessments or clinical tests while participating in this study will be captured. The study coordinator will contact participants virtually to answer questions and assess adverse effects after Titration period, Fixed-Dose period, and 4 weeks after Taper.

# Taper Down: maximum duration 2 weeks

Upon completion of the Fixed-Dose period, all participants in the study will be titrated off study drug through a taper down period of maximum 2 weeks. Taper schedule will directly relate to maximum gabapentin dose achieved during trial and is described in the Table below. The study drug will be distributed in 2 separate vials representing each of the two weeks of the Taper-Down Period. It should be noted, participants randomized to placebo will also receive sufficient capsules to complete a taper down. In this way, the blind will be maintained.

| AT 3600 MG | AT 2700 MG | AT 1800 MG | AT 900 MG |
|---|---|---|---|
| FOR 3 DAYS<br>3 MORNING<br>3 NOON<br>3 NIGHT | FOR 3 DAYS<br>2 MORNING<br>2 NOON<br>2 NIGHT | FOR 3 DAYS<br>1 MORNING<br>1 NOON<br>1 NIGHT<br>THEN STOP | NO TAPER<br>REQUIRED |
| NEXT 3 DAYS<br>2 MORNING<br>2 NOON<br>2 NIGHT | NEXT 3 DAYS<br>1 MORNING<br>1 NOON<br>1 NIGHT<br>THEN STOP | | |
| FINAL 3 DAYS<br>1 MORNING<br>1 NOON<br>1 NIGHT<br>THEN STOP | | | |

# Gabapentin Taper Down Schedule

End of Study Intervention: Exit Interview/ Data Collection: 4 weeks after completing Taper Down

The RA will contact the participants to query participants about compliance with taper-down schedule and maintenance of diaries. Participants will complete the following forms (survey titled: "FinalSurvey"):

- 1. Clinical Global Impression of Severity Scale (CGI-S).
- 2. Clinical Global Impression of Improvement Scale (CGI-I)
- 3. University of Pennsylvania Smell Identification Test (UPSIT)
- 4. Olfactory Dysfunction Outcomes Rating (ODOR)
- 5. NASAL-7
  - 6. Clinical Global Impression-Severity Scale for Parosmics (CGI-P)

# F3 Safety and Adverse Events

### 3.a Safety and Compliance Monitoring

- The specific monitoring plan for this study is based on the potential risk of participation and size and complexity of the planned investigation. Based on these considerations, this
- study will have a monitoring committee comprised of Dr. Piccirillo, Ms. Kukuljan, and
- Dr. Kallogjeri, the study biostatistician. All reports of a Serious Adverse Event (SAE) or

an Unexpected Adverse Event (UAE) will be investigated by the monitoring team and reported to Washington University HRPO according to the reporting requirements.

Participants who experience serious adverse effects with gabapentin therapy will be removed from the study. Participants with serious adverse effects will be instructed to call 911, seek immediate medical care and discontinue all further gabapentin treatment. If tolerated, all participants will complete the Titration period (≤ 4 weeks), Fixed-Dose period (8 weeks), and Taper-Down period (2 weeks) for maximum 14 weeks of active participation. In addition, there will be a 4-week, post-Taper completion follow-up for

maximum total of 18-week trial duration.

# 3.a Medical Monitoring

# i Investigator only

The PI and the study team will be monitoring patients for any safety concerns, such as SAE or UAE, in real time for the duration of the 18-week study. In addition, participants will be specifically asked about any adverse events after the Fixed-Dose period via REDCap. Participants will be able to get in touch with a member of the study team 24/7 via phone or pager for the duration of the 18-week clinical trial. The study biostatistician will hold the randomization codes and remain blinded to the intervention assignment. In the event of an SAE or UAE in which the blind needs to be broken, the Research Pharmacist will be contacted by the PI or a member of the study team. The participant will receive appropriate care and will be removed from the trial. A description of the event will be included in the report of adverse events for the clinical study.

#### 3.b Definitions of Adverse Events

Adverse event (AE) means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related (21 CFR 312.32(a)).

An adverse event (also referred to as an adverse experience) can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporarily associated with the use of a drug, without any judgment about causality or relationship to the drug.

An adverse event can arise from any use of the drug (e.g., off-label use, use in combination with another drug) and from any route of administration, formulation, or dose, including an overdose.

Serious adverse events (SAEs) are special cases of an adverse event where adverse outcomes are severe. SAEs include the following events:

- Death of any of the participants associated with a clinical trial.
- An event which can lead to life-threatening complications or put the life of participants at risk as a result of participation in a clinical trial.

- Events that result in such a condition where the participants may require immediate hospitalization or increase the duration of hospitalization.
  - Any events that lead to a permanent or temporary physical disability in the body of the participants. Any sort of incapacity is also regarded as SAE.
  - Any events that lead to any type of congenital abnormalities. It also includes any cases of birth defects resulting from the clinical trials.
  - Any events where an investigator or team of investigators finds feel that it can lead to significant hazards.

# **Classification of Events**

698

699

700

701 702

703

704

705

706 707

708

709

716

717

720

721

722

723 724

725

726

727

728

729

730

731

737

# i Relationship

- An AE or SAE may or may not be causally related to the study intervention. A causal
- relationship means that the intervention caused (or is reasonably likely to have caused)
- the AE. This usually implies a relationship in time between the intervention and the AE
- 713 (e.g., the AE occurred shortly after the participant received the intervention). For all
- AEs, it is the responsibility of the Principal Investigator who examines and evaluates the
- patient to determine the relatedness of the event to the study intervention.

# ii Severity

- Severity refers to the intensity of a specific event and is a matter of individual clinical judgment.
  - Grade 1: Asymptomatic or mild symptoms; clinical or diagnostic observations only; no intervention indicated
  - Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)
  - Grade 3: Severe; or medically significant but not immediately life- threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL
  - Grade 4: Life-threatening; urgent intervention indicated.
  - Grade 5: Death related to an AE

### iii Expectedness

- An adverse event or suspected adverse reaction is considered "unexpected" if it is not
- consistent with the risk information described in this protocol or on the informed consent
- or is not listed at the specificity or severity that has been observed; or, if an investigator
- brochure is not required or available, is not consistent with the risk information described
- in the general investigational plan or elsewhere in the current application, as amended.

### 3.c Data Collection Procedures for Adverse Events

- All adverse events and suspected adverse reactions are collected from 'source
- documentation' and the research coordinator will abstract the events. Documentation can

740 be within Washington University EPIC medical records, but at times the research

coordinator will also need to have the subject or family send outside source

742 documentation.

743

744

741

#### **3.d Reporting Procedures**

- The Principal Investigator (PI) will be responsible for ensuring participants' safety on a 745
- daily basis and for reporting Serious Adverse Events and Unanticipated Problems to the 746
- 747 Institutional Review Board (IRB) as required.

748

749 All SAEs will be reported immediately to the Principal Investigator upon identification.

#### 3.e **Adverse Event Reporting Period**

750 751

752 All AEs and unanticipated problems will be reported to the IRB in a prompt and timely

753 manner to protect other subjects from avoidable harm. The appropriate time frame for 754

satisfying the requirement for prompt reporting will vary depending on the specific nature

755 of the unanticipated problem. For this study, unanticipated problems that are serious

756 adverse events will be reported to the IRB within 1 week of the investigator becoming 757

aware of the event. Any other unanticipated problem will be reported to the IRB within 2

758 weeks of the investigator becoming aware of the problem.

759 760

Determining the appropriate time frame for reporting a particular unanticipated problem

761 requires careful judgment by the Research Coordinator and the Principal Investigator

762 knowledgeable about human subject protections. The primary consideration in making 763

these judgments is the need to take timely action to prevent avoidable harms to other subjects.

764

765

766

767

#### **F4** Study Outcome Measurements and Ascertainment

Participants will complete an assessment of blind after completion of 4 weeks of the 8-week Fixed-Dose period using REDCap (survey titled: "Blind Assessment")

768 769 770

Participants will also complete the following forms using REDCap (survey titled "FixedDoseSurvey") after completing the 8-week Fixed-Dose Period:

771 772 773

774

775

776

777

778

- 1.) Clinical Global Impression of Severity Scale (CGI-S).
- 2.) Clinical Global Impression of Improvement Scale (CGI-I)
- 3.) University of Pennsylvania Smell Identification Test (UPSIT)
  - 4.) Olfactory Dysfunction Outcomes Rating (ODOR)
  - 5.) *NASAL-7*
  - 6.) Clinical Global Impression-Severity Scale for Parosmics (CGI-P)
- 779 7.) Adverse Event assessment
- 780 8.) Compliance

782 Participants will also complete the following forms using REDCap (survey titled 783 FinalSurvey) 4 weeks after completing the Taper Period.

- 1) Clinical Global Impression of Severity Scale (CGI-S).
- 2) Clinical Global Impression of Improvement Scale (CGI-I)
- 3) University of Pennsylvania Smell Identification Test (UPSIT)
- 787 4) Olfactory Dysfunction Outcomes Rating (ODOR)
- 788 5) NASAL-7

**Statistical Plan** 

789 6) Clinical Global Impression-Severity Scale for Parosmics (CGI-P)

790

784

785

786

791

# 792

793

794

795

796

797

798

799

800

801

802

803

804

805

806

807

808

809

#### **G**1 Sample Size Determination and Power

To date there have been no studies investigating efficacy of gabapentin in COVID-19 related olfactory dysfunction. Due to the lack of preliminary data and effect size, estimates of the sample size for this study will be determined based on feasibility. For this pilot study, we plan to enroll 60 subjects. The sample size of 60 subjects is feasible given the incidence of COVID-19 cases in Missouri and considering a conservative estimate of a 10% rate of permanent olfactory dysfunction among those (~50%) who experience olfactory dysfunction as one of the presenting symptoms. Using a 33% drop out rate, we estimate that the sample size of 60 subjects randomized in a balanced way between the two treatment groups will provide us with 40 evaluable cases. A previous study exploring a different treatment for COVID-19 related anosmia in our lab showed that 30% of the participants randomized to placebo reported improvement at the end of the trial as compared to baseline. We aim to observe a 25% difference in the response rate between gabapentin and placebo groups. Assuming that this will be the response rate in the placebo group of our trial, the sample size of 20 subjects per group will provide us with a 95% Confidence Interval -5% to 55% around the desired proportion difference of 25% between gabapentin and placebo groups.

810 811

812

#### *G2* Interim Monitoring and Early Stopping

- 813 There will not be a planned interim monitoring, nor will there be early stopping rules.
- 814 Statistical Methods **G**3
- 815 An intention-to-treat analysis will be used for the primary analysis of the data. All
- 816 participants will be examined in the groups to which they were initially assigned.
- 817 Standard descriptive statistics will be used to assess the demographics, clinical
- 818 characteristics, and olfactory test results of the study population. The difference in rate of
- 819 responders after Fixed-Dose period will estimate the effect size of the primary outcome
- 820 measure, and the 95% CI around that point estimate will measure precision. In each
- 821 group, the frequency and relative frequency of the participants' response to the global
- 822 rating of smell change will be reported for each Likert category. Fisher's exact test will
- 823 be used for comparing the responders' rates between the 2 groups. Histograms and

824 Shapiro-Wilks test will be used to test the normal distribution assumption of the 825 continuously measured UPSIT scores and the differences pre-post treatment in each of 826 the groups. Independent samples t-test or its nonparametric equivalent Mann-Whitney U 827 test will be used to compare the change in UPSIT scores between the two groups. Mixed 828 effects model will be used to test whether the change in UPSIT score from baseline to 829 end of treatment is significantly different between 2 groups. Subjects will be treated as 830 random factors, and group and time will be used as fixed factors in the model. Interaction 831 of group by time will be explored. Effect sizes with 95% CIs will be reported for each

832 analysis. All statistical analyses will be conducted in SPSS 28 (IBM Corp., Armonk, 833 NY).

834

835

840

841 842

#### **G**4 Missing Outcome Data

- 836 All attempts will be made using Good Clinical Practice and through the reduction of the 837 complexity and number of assessments to minimize the occurrence of missing outcome 838 data. It will be assumed that all missing data will be at random. As this is a small pilot
- 839 study, no computational techniques will be employed to adjust analyses for missing data.

#### **Unblinding Procedures G**5

- The blind will be broken for individual participants for safety concerns. Knowledge of the treatment received is necessary for interpreting the event, may be essential for the
- 843 medical management of the subject, and may provide critical safety information about
- 844 gabapentin that could have implications for the ongoing conduct of the trial (e.g.,
- 845 monitoring, informed consent). For unblinding, the research coordinator will contact the
- 846 research pharmacist and provide the study ID number for the participant to be unblinded.
- 847 The research pharmacist will contact the PI directly and reveal the intervention 848 assignment. The research coordinator will remain blinded.

849

### **Data Handling and Record Keeping**

851

852

850

#### *H1* Confidentiality and Security

- 853 Procedures that are in place to curb risks of breaches in confidentiality and privacy are 1) 854 formal training protocols centered on the maintenance of confidentiality for all study team members and secure storage for identified data such as completed questionnaires 855
- 856 and UPSIT exams; and communication with study team via secure email, phone line, or
- 857 televideo call.

858 859

860

861

862

863

Only members of the study team will have access to the electronic research files. All research data files will be stored on secure Washington University servers with computer, network, and database-level passwords that will only be accessible to study team members. Accordingly, these mechanisms intend to limit access to information that can link clinical data to individual participants. No participant identifying information will be revealed in any publications or presentations.

866 Case report forms will be created as electronic documents and stored within each study 867 participants electronic file. Original hard-copy source documents will be electronically scanned and stored in the participants electronic file and stored in a locked file cabinet. 868 869 H2**Records Retention** 870 All records will be retained for a minimum of six years after completion of the study and 871 closure with the WU IRB. 872 **Study Administration** 873 874 **I1** Subject Stipends or Payments 875 Participants will be provided a Forte/Advarra debit card. They will receive \$60 for 876 completing all study requirements. If participants do not complete all requirements, they 877 will be paid proportionally for the work they have completed. 878 879 *I2* Study Timetable 880 881 January 2022: IRB approval process and acquisition of resources 882 February 2022 - March 2022: Rolling recruitment 883 February 2022 - August 2022: 18-week clinical trial 884 September 2022: Statistical analysis and publication of results 885 886 J **Publication Plan** 887 888 We plan to analyze accumulated data throughout the month of September 2022 and 889 publish the results by the end of September 2022. This data includes the analysis of the 890 CGI-I, UPSIT, ODOR, NASAL-7, and CGI-P as well as a discussion of the potential 891 adverse effects associated with oral gabapentin therapy for treatment of post-COVID-19 892 olfactory dysfunction. 893 894 K **Attachments** 895 *K1* Questionnaires or surveys 896 Screening Survey 897 Screening UPSIT 898 Week0BaselineSurvey 899 Blind Assessment 900 FixedDoseSurvey 901 FinalSurvey 902 903

### L References

905 906

- 907 1. Prevention CfDCa. COVID Data Tracker. <a href="https://covid.cdc.gov/covid-data-tracker/#datatracker-home">https://covid.cdc.gov/covid-data-tracker/#datatracker-home</a>. Published 2021. Accessed.
- Organization WH. WHO Coronavirus (COVID-19) Dashboard.
   <a href="https://covid19.who.int/">https://covid19.who.int/</a>. Published 2021. Accessed.
- 911 3. Lechien JR, Chiesa-Estomba CM, De Siati DR, et al. Olfactory and gustatory 912 dysfunctions as a clinical presentation of mild-to-moderate forms of the 913 coronavirus disease (COVID-19): a multicenter European study. *Eur Arch* 914 *Otorhinolaryngol*. 2020.
- 915 4. Boscolo-Rizzo P, Borsetto D, Fabbris C, et al. Evolution of Altered Sense of
   916 Smell or Taste in Patients With Mildly Symptomatic COVID-19. *JAMA* 917 Otolaryngol Head Neck Surg. 2020.
- Hummel T, Rissom K, Reden J, Hahner A, Weidenbecher M, Huttenbrink KB.
   Effects of olfactory training in patients with olfactory loss. *Laryngoscope*.
   2009;119(3):496-499.
- 921 6. Turner JH. Olfactory training: what is the evidence? *Int Forum Allergy Rhinol*. 2020;10(11):1199-1200.
- Biole C, Bianco M, Nunez-Gil IJ, et al. Gender Differences in the Presentation
   and Outcomes of Hospitalized Patients With COVID-19. *J Hosp Med*.
   2021;16(6):349-352.
- 926 8. Butowt R, von Bartheld CS. Anosmia in COVID-19: Underlying Mechanisms and
   927 Assessment of an Olfactory Route to Brain Infection. *Neuroscientist*.
   928 2020:1073858420956905.
- 929 9. Bilinska K, Butowt R. Anosmia in COVID-19: A Bumpy Road to Establishing a Cellular Mechanism. *ACS Chem Neurosci.* 2020;11(15):2152-2155.
- 931 10. Kuba K, Imai Y, Penninger JM. Multiple functions of angiotensin-converting 932 enzyme 2 and its relevance in cardiovascular diseases. *Circ J.* 2013;77(2):301-933 308.
- 934 11. Mollica V, Rizzo A, Massari F. The pivotal role of TMPRSS2 in coronavirus disease 2019 and prostate cancer. *Future Oncol.* 2020;16(27):2029-2033.
- Damm M, Pikart LK, Reimann H, et al. Olfactory training is helpful in postinfectious olfactory loss: a randomized, controlled, multicenter study.
   *Laryngoscope*. 2014;124(4):826-831.
- 939 13. Schopf CL, Ablinger C, Geisler SM, et al. Presynaptic alpha2delta subunits are key organizers of glutamatergic synapses. *Proc Natl Acad Sci U S A*. 941 2021:118(14).
- 942 14. Lopez-D'alessandro E, Escovich L. Combination of alpha lipoic acid and gabapentin, its efficacy in the treatment of Burning Mouth Syndrome: a randomized, double-blind, placebo controlled trial. *Med Oral Patol Oral Cir Bucal.* 2011;16(5):e635-640.
- Doty RL, Shaman P, Dann M. Development of the University of Pennsylvania
   Smell Identification Test: A standardized microencapsulated test of olfactory
   function. *Physiol Behav*. 1984;32(3):489-502.

- 949 16. Doty RL. Olfactory dysfunction and its measurement in the clinic. *World J Otorhinolaryngol Head Neck Surg.* 2015;1(1):28-33.
- 951 17. Mersfelder TL, Nichols WH. Gabapentin: Abuse, Dependence, and Withdrawal. 952 Ann Pharmacother. 2016;50(3):229-233.